CLINICAL TRIAL: NCT05919420
Title: White-coat Hypertension in Childhood - Effects on Blood Pressure and Organ Damage
Acronym: WCH
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Rafael T Krmar, MD PhD, Medical doctor, PhD, Karolinska Institutet
Other Study IDs: WCH
Record Dates: First submitted 2015-12-09; First posted 2023-06-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-06

CONDITIONS: White Coat Hypertension
MeSH Terms: conditions — White Coat Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
White coat hypertension, WCH means that the blood pressure are above normal values only when measured at visits to the doctor, but not at home. WCH has in adults proved to be predisposing to the development of hypertension, and damage to the heart and arteries. It is not known if children and young people run the same risk as adults with WCH.

The investigators have previously examined the blood pressure of 1473 healthy children and adolescents in the study "Screening for high blood pressure and silent kidney disease in school children" and the results were published recently in the American Journal of Hypertension. In the study, we identified a number of participants who had the WCH.

The investigators are implementing now, 10 years later, a follow-up study to investigate if these children with WCH have an increased risk of hypertension and subsequent cardiovascular disease. The goal is to investigate whether these young individuals are at similar risk as adults with WCH for hypertension and impaired cardiovascular function.

The investigators will provide our WCH participants extended examinations of the heart, blood vessels and kidney function, which will provide important information as to whether there are effects on cardiovascular health already in adolescence among participants that suffered from WCH in childhood. This is important knowledge in clinical work in order to learn how to best care for these children to minimize their risk of future disease.

DETAILED DESCRIPTION:
This is a longitudinal study in which all patients with WCH who previously participated in the above-mentioned study are included. The PI will offer the participants an outpatient check-up, which means:

* measurement of blood pressure with ambulatory blood pressure measurement during 24 hours to study blood pressure level and variation in blood pressure during the day.
* ultrasound examination of the structure and function of the heart
* ultrasound examination of blood vessels for calculation of intima-media thickness
* investigation of vessel elasticity with pulse wave analysis with Arteriograph.
* analysis of blood and urine to examine kidney function.
* Questionnaire about eating habits and physical activity

These examinations will be carried out at the Physiology Clinic, Karolinska University Hospital, Huddinge. Both ultrasound examination of blood vessels and pulse wave velocity are non-invasive examinations and provide important information about the patient's vascular status. We will take a venous blood sample (approx. 5 ml) for analysis of standard markers for organ damage and vascular function (creatinine, urate, urea, cystatin C) and a urine sample (urine albumin/creatinine). These standard measurements and sampling involve a minimal impact on the individual and the subsequent analysis methods are well developed and have been applied in several previous studies. We will also ask questions about lifestyle, which is part of the doctor's medical history. In cases where hypertension, with or without organ damage, is verified, the persons will be referred further to pediatric nephrology or to adult medicine.

The sampling is recorded according to usual routines and the participation in the study is also indicated.

Each participant is assigned a code number. Some patient-related clinical data will be recorded, such as body measurements and analysis results from blood sampling. Questionnaire responses and results from examinations from cardiac echocardiography, vascular doppler and pulse wave velocity are coded. The code list is kept separately in a locked space. Participating researchers all have access to the code list. During data processing, only coded information is used.

ELIGIBILITY:
Inclusion Criteria:

* being identified in our previous study as having WCH

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 56 participants with WCH that were identified in a previous study
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Hypertension | at follow up (average 9,3 years after baseline)
  blood pressure at hypertensive level
Left ventricular hypertrophy | at follow up (average 9,3 years after baseline)
  echocardiographic measurment
vascular elasticity | at follow up (average 9,3 years after baseline)
  pulse wave velocity